CLINICAL TRIAL: NCT05793151
Title: A Stepped Wedge Cluster Randomized Trial Comparing a Navigation-Based Multilevel Intervention With Treatment as Usual to Improve Initiation of Timely Postoperative Radiation Therapy in Adults With Head and Neck Cancer
Brief Title: Multi-Site Trial of Navigation vs Treatment as Usual to Improve Initiation of Timely Adjuvant Therapy
Acronym: ENDURE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Evan Graboyes, Associate Professor-Faculty, Medical University of South Carolina
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00123953; R01CA282165 (NIH)
Record Dates: First submitted 2023-03-20; First posted 2023-03-31 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Head and Neck Cancer; Head and Neck Squamous Cell Carcinoma; Oropharynx Cancer; Oral Cavity Cancer; Larynx Cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck; Oropharyngeal Neoplasms; Mouth Neoplasms; Laryngeal Neoplasms

STUDY DESIGN:
Intervention Model Description: Stepped Wedge Cluster Randomization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ENDURE (Experimental): ENDURE is a theoretically-informed, navigation-based, multilevel intervention targeting barriers to timely, guideline-adherent PORT.
  Interventions: Behavioral: ENDURE
- Treatment As Usual (No Intervention): Treatment as usual at each site consists of standard of care clinical practices

INTERVENTIONS:
Behavioral: ENDURE — ENDURE provides patient education through the ENDURE Patient Resource Guide and social support by linking patients to community resources (patient-level), standardizes discussions about expectations for PORT and clinical documentation to enhance communication and care coordination within and across interprofessional cancer teams (team-level), and implements referral tracking across fragmented health systems (organization-level). To facilitate care coordination, ENDURE modifies existing standard of care patient navigation (an evidence-based intervention that addresses barriers to timely cancer care) by adding PORT-focused navigation at three key care transitions: into the cancer care system; from inpatient to outpatient after surgery; and from the surgical team to the radiation oncology team.
  Arms: ENDURE

SUMMARY:
The goal of this clinical trial is to compare the effectiveness of a navigation-based multilevel intervention (ENDURE) with treatment as usual (TAU) to improve the initiation of guideline-adherent postoperative radiation therapy among patients with head and neck cancer. The main questions the trial aims to answer are:

1. Does ENDURE improve initiation of timely PORT relative to treatment as usual?
2. What are the mechanisms through which ENDURE improves timeliness to treatment?
3. What are the barriers and facilitators to the implementation of ENDURE into routine clinical care?

DETAILED DESCRIPTION:
In this hybrid type 1 effectiveness-implementation study, the investigators will conduct a stepped-wedge cluster randomized trial with cancer centers (n=4; 484 patients) randomized to sequentially deliver treatment as usual (TAU) then ENDURE to patients with head and neck cancer undergoing surgery and postoperative radiation therapy (PORT). The trial will assess the effect of ENDURE vs TAU on improving initiation of timely PORT (primary objective) and the underlying mechanisms of ENDURE (secondary objective). The investigators will concurrently conduct a mixed-methods study with quantitative measures of implementation outcomes and qualitative data about implementation determinants from semi-structured interviews with key stakeholders and site visits (exploratory objective).

ELIGIBILITY:
Inclusion Criteria:

1. Age >/= 18 years
2. Squamous cell carcinoma (SCC) (or histologic variant) of the oral cavity, oropharynx, hypopharynx, larynx, unknown primary, paranasal sinuses, or nasal cavity
3. American Joint Committee on Cancer (AJCC) 8th edition clinical T3-4 or >N1 SCC of the oral cavity, oropharynx, hypopharynx, larynx, paranasal sinuses, nasal cavity, or unknown primary.
4. No history of radiation therapy for treatment of HNSCC in the definitive or adjuvant settings that would, at the discretion of the enrolling clinician, affect the patient's need for adjuvant RT.
5. Plan for curative intent surgery at one of the participating centers
6. Plan for PORT (regardless of whether it is at the surgical center) with or without concurrent chemotherapy following curative intent surgery based on the expectation of at least one of the following adverse features on final pathologic evaluation: pT3 or pT4 primary, N1 or greater nodal disease, perineural invasion (PNI), or lymphovascular invasion (LVI).

Exclusion Criteria:

1. Inability to speak or read English or Spanish.
2. Severe mental illness that would prevent trial participation.
3. HPV-positive OPC or unknown primary SCC staged as cT1-2N1 with a single ipsilateral LN < 3 cm
4. Synchronous untreated malignancy expected to impact life expectancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 532 (Estimated)
Dates: Start 2023-10-30 (Actual); Primary Completion 2028-03-30 (Estimated); Study Completion 2028-03-30 (Estimated)

PRIMARY OUTCOMES:
Initiation of Timely PORT | 3 months
  The initiation of PORT > 6 weeks (42 days) following definitive surgery for HNSCC.

SECONDARY OUTCOMES:
Time-to-PORT | 4 months
  The number of days from the date of definitive surgery for HNSCC to the date of initiation of PORT.
Pre-Surgical consultation with radiation oncology | 1 month
  Consultation with a treating radiation oncologist prior to definitive surgery for HNSCC.
Pre-radiation therapy dental extractions | 1 month
  The removal of indicated carious/non-restorable teeth prior to or during the surgery for HNSCC.
Time to postoperative scheduling with radiation oncology | 3 months
  The time from definitive surgery to the placement of the postoperative referral (or follow-up appointment) with the treating radiation oncologist.
Time to postoperative appointment with radiation oncology | 3 months
  Time from definitive surgery to the attendance at an appointment with the treating radiation oncologist.

CONTACTS AND LOCATIONS:
Overall Officials: Evan M Graboyes, MD, MPH, Principal Investigator — Medical University of South Carolina
Locations (4):
- United States (4):
  - Washington University in St. Louis, St Louis, Missouri
  - Duke University Medical Center, Durham, North Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
Below are the key elements of the data sharing plan as outlined in the NIH Policy for Data Management and Sharing:
  Research materials will include: (1) self-report measures from patients; (2) clinical data from the electronic medical record; (3) audio recordings and transcriptions of interviews from stakeholders; and (4) field notes from direct observations of the delivery of ENDURE at each site. Data will be raw or minimally processed. The investigators plan to use REDCap for data capture and management of the clinical and self-report measure data and NVivo for management of the qualitative data. REDCap data dictionaries can be distributed for reuse. The final data dictionaries have not been developed. Scientific data and metadata will be generated, preserved, and shared using NIH common data elements. Scientific data and metadata arising from the project will be uploaded to openICPSR, a self-publishing repository for social, behavioral, and health sciences research data.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be shared no later than the time of a publication of findings of the trial's primary endpoint in a peer-reviewed journal.
Access Criteria: All data sharing will comply with privacy and confidentiality protections such as the NIH Certificate of Confidentiality and applicable laws, regulations, and policies governing data derived from human participants.